CLINICAL TRIAL: NCT01843387
Title: A Randomized, Controlled, Dose-Escalation Pilot Study to Assess the Safety and Efficacy of a Single Intravenous Infusion of Allogeneic Mesenchymal Precursor Cells (MPCs) in Subjects With Diabetic Nephropathy and Type 2 Diabetes
Brief Title: Safety and Efficacy of Mesenchymal Precursor Cells in Diabetic Nephropathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mesoblast, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MSB-DN001
Record Dates: First submitted 2013-04-23; First posted 2013-04-30 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Diabetic Nephropathy; Type 2 Diabetes
Keywords: Diabetic nephropathy; Chronic kidney disease; Metabolic disease; Diabetes mellitus, type 2
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic; Metabolic Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Experimental): Mesenchymal Precursor Cells (MPCs) - Dose 1 or Placebo
  Interventions: Biological: Mesenchymal Precursor Cells (MPCs)
- Cohort 2 (Experimental): Mesenchymal Precursor Cells (MPCs) - Dose 2 or Placebo
  Interventions: Biological: Mesenchymal Precursor Cells (MPCs)

INTERVENTIONS:
Biological: Mesenchymal Precursor Cells (MPCs) — Single Intravenous Infusion of MPCs Dose 1 or Placebo
  Arms: Cohort 1
Biological: Mesenchymal Precursor Cells (MPCs) — Single Intravenous Infusion of MPCs Dose 2 or Placebo
  Arms: Cohort 2

SUMMARY:
The study investigates the safety, tolerability and efficacy of a single intravenous infusion of two doses of mesenchymal precursor cells versus placebo in subjects with diabetic nephropathy and type 2 diabetes.

DETAILED DESCRIPTION:
This study is taking place in Melbourne, Australia.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who are ≥ 50 and ≤ 85 years old
* Subjects diagnosed with type 2 diabetes at least 2 years prior to Screening
* Subjects with diabetic nephropathy and CKD stage 3b-4
* Albumin-to-creatinine ratio (ACR) from a spot urine sample >30 and < 3000 mg/g at Screening
* Subjects must be receiving standard of care treatment for their diabetic nephropathy with an angiotensin converting enzyme inhibitor (ACEi) and/or an angiotensin II receptor blocker (ARB) for at least 12 weeks prior to Screening.
* HbA1c < 10.0% at Screening

Exclusion Criteria:

* Prior participation in any stem cell study
* Women of childbearing potential
* Potentially unreliable subjects and those judged by the Investigator to be unsuitable for the study
* History of active substance abuse (including alcohol) within the past 2 years. Current alcohol abuse is defined as daily consumption of >3 alcoholic beverages (i.e. > 21 alcoholic beverages per week)
* Body weight >150 kg
* Subjects with non-diabetic renal disease e.g. known polycystic kidney disease
* Subjects with a history of a renal transplant or who have had prior dialysis within 3 months of Screening and/or have not maintained a stable level of kidney function within 3 months of Screening
* Current or history within 6 months of Screening of NYHA Class III or IV heart failure
* Myocardial infarction or stroke within 6 months prior to Screening
* Any concurrent medical condition/disorder or clinically symptomatic cardiovascular, gastrointestinal, hematological, pulmonary, acute or chronic infectious disease, active retinal disease or other disorder which in the Investigator's opinion would interfere with the subjects ability to complete the trial, would require administration of treatment that could affect the interpretation of the efficacy and safety variables or would preclude safe involvement in the study

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-07; Primary Completion 2014-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to assess the safety and tolerability of MPC therapy | 60 Weeks
  Outcomes include the following safety parameters:
  * Number of and percent of subject with adverse events and serious adverse events
  * Clinically significant values and shifts from baseline in vital signs, physical examinations and electrocardiograms
  * Clinical laboratory tests (hematology, chemistry and urinalysis, flow cytometry with Class I and Class II PRA % with specificity)

SECONDARY OUTCOMES:
Exploratory assessment of the efficacy of MPC therapy | 12 Weeks
  Outcomes include changes from baseline at 12 weeks in the following parameters:
  * Renal function (glomerular filtration rate, renal blood flow)
  * Serum creatinine
  * Urinary albumin and protein excretion
  * Glycemic control
  * Biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: K Segal, PhD, Study Director — Mesoblast, Ltd.
Locations (2):
- Australia (2):
  - Monash Universtiy, Clayton
  - Melbourne Renal Research Group, Melbourne

REFERENCES:
- [Derived] Packham DK, Fraser IR, Kerr PG, Segal KR. Allogeneic Mesenchymal Precursor Cells (MPC) in Diabetic Nephropathy: A Randomized, Placebo-controlled, Dose Escalation Study. EBioMedicine. 2016 Oct;12:263-269. doi: 10.1016/j.ebiom.2016.09.011. Epub 2016 Sep 17. PMID 27743903